CLINICAL TRIAL: NCT00941785
Title: Randomized Trial of the Efficacy, Safety, Tolerability and Pharmacokinetics of Dihydroartemisinin-piperaquine for Seasonal IPT to Prevent Malaria in Children Under 5 Years
Brief Title: Dihydroartemisinin (DHA)-Piperaquine for IPT to Prevent Malaria in Children in Burkina Faso
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: BEIJING HOLLEY-COTEC PHARMACEUTICALS CO. LTD. (Unknown)
Responsible Party: Dr Issaka Zongo, IRSS, BP 545 Bobo-Dioulasso (Burkina Faso)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC5550
Record Dates: First submitted 2009-06-18; First posted 2009-07-20 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Malaria
Keywords: Malaria; Intermittent Preventive Treatment; IPTc; sIPTc; Burkina Faso
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA-PQ (Experimental): Three monthly administrations of dihydroartemisinin (DHA) plus piperaquine (PQ) in August, September and October.
  Interventions: Drug: DHA-PQ
- SP-AQ (Active Comparator): Three monthly administrations of sulfadoxine-pyrimethamine plus amodiaquine
  Interventions: Drug: SP-AQ

INTERVENTIONS:
Drug: DHA-PQ — Three monthly administrations of Duocotexcin (DHA-PQ):
  dihydroartemisinin 2.1mg/kg and piperaquine phosphate 16.8 mg/kg once daily for three days
  Other Names: Seasonal IPTc with Duocotexcin (Holley)
  Arms: DHA-PQ
Drug: SP-AQ — Three monthly administrations of sulfadoxine-pyrimethamine plus amodiaquine:
  One dose of Sulfadoxine 25mg/kg and pyrimethamine 1.25mg/kg Three daily doses of amodiaquine phosphate 10mg/kg
  Other Names: Seasonal IPTc with Fansidar plus amodiaquine (Flavoquine)
  Arms: SP-AQ

SUMMARY:
The aim of the study is to determine whether piperaquine plus dihydroartemisinin (DHA-PQ) is as effective, and better tolerated, than sulfadoxine-pyrimethamine plus amodiaquine (SP+AQ), when used for seasonal Intermittent Preventive Treatment (IPT) to prevent malaria in children aged 3 to 59 months in Bobo-Dioulasso, Burkina Faso and to determine the pharmacokinetics of piperaquine in children.

DETAILED DESCRIPTION:
There is evidence from several studies that in areas where the transmission of malaria is seasonal, the use of IPT can reduce substantially the incidence of clinical malaria in children under the age of five years, by as much as 90% (Greenwood et al, Trends in Parasitology 24(11):485-6, 2008). The most effective regimen is SP+AQ but alternative regimens are needed because amodiaquine can be poorly tolerated (Sokhna et al PlosOne 3:e1471, 2008) and resistance to SP is increasing. In recent trials in Senegal and The Gambia, PQ combined with DHA or SP was as effective against malaria, and better tolerated, than SP+AQ. Of these regimens, only DHA+PQ is licensed for use as an antimalarial in African countries. However there are no data on pharmacokinetics of PQ when used for IPT in children, and the impact of DHA+PQ in preventing spread of resistance is not known. This trial aims to provide this information in order to evaluate the suitability of DHA+PQ for use for seasonal IPT in children and to determine the optimum dose regimen for piperaquine.

Malaria (caused primarily by Plasmodium falciparum) is endemic in the southern third of Burkina Faso, occurring seasonally between June to November, with most cases occurring between August and October. In Burkina Faso there has been no evidence of a recent decline in malaria incidence as seen in some other African countries. Although the policy is to treat uncomplicated malaria with artemisin combinations, in practice chloroquine remains the treatment used in most health facilities. Several studies have shown that seasonal IPT in children (IPTc) can provide a high degree of protection against clinical malaria. SP+AQ is the most effective regimen but amodiaquine is not well tolerated and resistance to SP is increasing n many areas. Alternative regimens are required. Piperaquine (PQ), a long acting antimalarial used for prophylaxis in China, is suitable for use for IPT. In studies in Senegal and The Gambia piperaquine plus SP or dihydroartemisinin (DHA) was as effective and better tolerated than SP+AQ. The purpose of this study is to determine whether DHA-PQ is more effective than SP+AQ in preventing spread of drug resistant parasite genotypes and to determine the pharmacokinetics of piperaquine in children who receive this drug for IPT. Little was known about the pharmacokinetics of piperaquine until recently, and there is currently only limited information about the pharmacokinetics of piperaquine in children. The pharmacokinetic data from this study will allow us to estimate the optimum dose regimen for piperaquine; the current recommended regimen for DHA-PQ is three doses over three days. For IPT, a single dose regimen is highly desirable as it would be easier to deliver and better accepted by communities.

1500 children aged 3 to 59 months will be enrolled and randomized to receive 3 monthly administrations of DHA-PQ or SP-AQ, in August, September and October. From August to November children will be visited twice weekly to check for malaria symptoms.

A subset of 45 children in each treatment group will be asked to provide a venous blood sample on days 0 and 7 for analysis of biochemical and haematological parameters.

In the DHA-PQ group only, a subset of 210 children will be asked to provide finger prick blood samples for PK analysis on day 0, between day 0 and day 6, on day 7, and between day 8 and day 30. To calibrate measurements of drug concentration in peripheral blood against existing PK models, each month 17 of these children will be asked to also provide a venous sample (up to 2ml taken into a vacutainer) on three occasions (one between day 0 and 6, one on day 7, and one between day 8 and 30). In addition, a separate group of 750 children aged 3 to 59 months will be recruited to be surveyed at the end of the transmission season to determine the prevalence of malaria parasitaemia and of drug-resistance parasite genotypes in the study area.

ELIGIBILITY:
Inclusion Criteria:

* signed consent from a parent
* age 3-59 months at enrolment
* no history of allergy to study drugs
* no chronic illness

Exclusion Criteria:

* history of allergy to study drugs
* intention to move away from the study area before the end of 2009
* any chronic illness

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Efficacy against clinical malaria | August to December 2009
Incidence of adverse events | Within 7 days of each treatment round and within 1 month of treatment

SECONDARY OUTCOMES:
Pharmacokinetics of piperaquie: the oral clearance (CL/F), AUC, steady state volume of distribution(s) (Vss/F), inter-compartment clearance(s) (Q/F) and absorption rate (ka) will be estimated. | during 30 days after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bosco Ouédraogo, MD, Study Director — IRSS, Direction Régionale,BP 545 Bobo-Dioulasso (Burkina Faso); Paul JM Milligan, PhD, Study Chair — London School of Hygiene and Tropical Medicine; Issaka Zongo, MD, Principal Investigator — IRSS, Burkina Faso and LSHTM, UK
Locations (1):
- IRSS, Bobo-Dioulasso, Bobo-Dioulasso, Burkina Faso

REFERENCES:
- [Derived] Zongo I, Milligan P, Compaore YD, Some AF, Greenwood B, Tarning J, Rosenthal PJ, Sutherland C, Nosten F, Ouedraogo JB. Randomized Noninferiority Trial of Dihydroartemisinin-Piperaquine Compared with Sulfadoxine-Pyrimethamine plus Amodiaquine for Seasonal Malaria Chemoprevention in Burkina Faso. Antimicrob Agents Chemother. 2015 Aug;59(8):4387-96. doi: 10.1128/AAC.04923-14. Epub 2015 Apr 27. PMID 25918149
- [Derived] Some AF, Zongo I, Compaore YD, Sakande S, Nosten F, Ouedraogo JB, Rosenthal PJ. Selection of drug resistance-mediating Plasmodium falciparum genetic polymorphisms by seasonal malaria chemoprevention in Burkina Faso. Antimicrob Agents Chemother. 2014 Jul;58(7):3660-5. doi: 10.1128/AAC.02406-14. Epub 2014 Apr 14. PMID 24733476